CLINICAL TRIAL: NCT00835731
Title: Cervical Preparation Before Same-day Second Trimester Abortion With Buccal Misoprostol Versus Dilapan-S: A Randomized Placebo Controlled Trial
Brief Title: Misoprostol Versus Dilapan-S for Cervical Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SFP2-3
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Cervical Ripening
Keywords: induced abortion; misoprostol; cervical ripening; second trimester abortion; Dilapan-S
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 400mcg buccal misoprostol
  Interventions: Drug: misoprostol
- 2 (Experimental): Dilapan-S, control: vitamin B-12 administered sublingually
  Interventions: Device: Dilapan-S, vitamin B-12

INTERVENTIONS:
Drug: misoprostol — 400mcg misoprostol, buccal administration, 1 time dosing 3-4 hours before abortion by D&E
  Other Names: Cytotec
  Arms: 1
Device: Dilapan-S, vitamin B-12 — One Dilapan-S rod placed in the cervix 3-4 hours before abortion by D&E. Control: 1000mcg vitamin B-12, buccal administration 3-4 hours before abortion by D&E
  Arms: 2

SUMMARY:
The purpose of this study is to compare the dilatory effect of 400 mcg of buccally administered misoprostol to one Dilapan-S rod placed 3-4 hours before abortion by dilation and evacuation in women who are 12 weeks 0 days to 15 weeks 0 days gestation.

ELIGIBILITY:
Inclusion Criteria:

* medically eligible for dilation and evacuation at Planned Parenthood League of Massachusetts
* gestational age 12 weeks 0 days to 15 weeks 0 days as evaluated by ultrasound
* proficient in English or Spanish
* agreeing to study procedures, including randomization and surveys regarding demographics, medical and gynecological history, and assessments of pain and satisfaction

Exclusion Criteria:

* less than 18 years old
* cervical or uterine anomaly that the research physician deems may affect the difficulty of dilation or the abortion procedure
* inflammatory bowel disease
* contraindication to misoprostol use
* known intolerance or allergy to misoprostol or Dilapan-S
* inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prinicpal Investigator, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352
- [Derived] Bartz D, Maurer R, Allen RH, Fortin J, Kuang B, Goldberg AB. Buccal misoprostol compared with synthetic osmotic cervical dilator before surgical abortion: a randomized controlled trial. Obstet Gynecol. 2013 Jul;122(1):57-63. doi: 10.1097/AOG.0b013e3182983889. PMID 23743471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: January 2009 - December 2011 We recruited English- or Spanish-speaking women who were in good health, at least 18 years old, and between 12 weeks 0 days and 15 weeks 0 days gestation by ultrasound examination, seeking outpatient pregnancy termination at Planned Parenthood League of MA.
Pre-assignment Details: Patients were recruited for study participation on the day of their pregnancy termination procedure. All study procedures occurred on the day that the patient was enrolled.
Groups:
- Misoprostol: 400mcg buccal misoprostol
  misoprostol : 400mcg misoprostol, buccal administration, 1 time dosing 3-4 hours before abortion by D&E
- Synthetic Osmotic Dilator: Dilapan-S, control: vitamin B-12 administered sublingually
  Dilapan-S, vitamin B-12 : One Dilapan-S rod placed in the cervix 3-4 hours before abortion by D&E.
  Control: 1000mcg vitamin B-12, buccal administration 3-4 hours before abortion by D&E
Period: Overall Study
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Started | 64 | 61
Completed | 62 | 60
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Synthetic Osmotic Dilator | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 61 | 125
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (5.5) | 24.0 (5.0) | 24.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 125
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cervical Dilation in Women Following Exposure to Either Ripening Agent
Time Frame: 3-4 hours after placement of ripening agent
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
mm | 32.1 (6.0) | 33.9 (4.7)

2. Secondary Outcome: Ease of Further Mechanical Dilation in Women Following Exposure to Either Ripening Agent, as Per MD Report
Description: Scale:
  None needed (score of 0) Very easy (score 1) Somewhat easy (score of 2) Moderate (score of 3) Somewhat difficult (score of 4) Very difficult (score of 5)
Time Frame: 3-4 hours after placement of ripening agent
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
Participants
  None needed (score of 0) | 3 | 3
  Very-somewhat easy (score of 1-2) | 29 | 27
  Moderate (score of 3) | 12 | 24
  Somewhat-very difficult (score of 4-5) | 18 | 6

3. Secondary Outcome: Procedure Time for Dilation and Evacuation
Time Frame: 3-4 hours after placement of ripening agent
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
minutes | 2.8 [2.0 to 3.8] | 3.0 [2.2 to 3.9]

4. Secondary Outcome: Number of Patients for Whom Physician Was Able to Complete Dilation and Evacuation Procedure on First Attempt
Time Frame: 3-4 hours after placement of ripening agent
Measure: Number; unit: participants
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
participants | 62 | 60

5. Secondary Outcome: Subject Pain During Ripening
Description: Measure assesses patient pain during cervical preparation. Pain was assessed after cervical ripening was complete, immediately before D&E procedure. Subjects were asked to rate pain on a 6 point Likert scale:
  0 = no pain 1-2 = mild pain 3 = moderate pain 4-5 = severe pain
  Higher values represent a worse outcome.
Time Frame: 3-4 hours after placement of ripening agent
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
Scores on a scale | 1 [1 to 3] | 1 [0 to 2]

6. Secondary Outcome: Subject Pain During Dilation and Evacuation
Description: Measure assesses subject pain during dilation and evacuation. Pain was assessed immediately after the D&E procedure. Subjects were asked to rate pain on a 6 point Likert scale:
  0 = no pain 1-2 = mild pain 3 = moderate pain 4-5 = severe pain
  Higher values represent a worse outcome.
Time Frame: 3-4 hours after placement of ripening agent
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
Scores on a scale | 3 [1 to 4] | 3 [1 to 4]

7. Secondary Outcome: Women's Satisfaction With Cervical Ripening Method
Description: Scale:
  1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, 5 = very satisfied
Time Frame: 5 hours after placement of ripening agent
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Number analyzed (Participants) | 62 | 60
units on a scale | 4 [3 to 5] | 4 [4 to 5]

ADVERSE EVENTS:
Arm/Group | Misoprostol | Synthetic Osmotic Dilator
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 3/62 | 3/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol (N=62) | Synthetic Osmotic Dilator (N=60)
Same-day re-evacuation (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) — estimated blood loss of 300 cc
Cervical laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) — minor, treated with cervical pressure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No